CLINICAL TRIAL: NCT06001866
Title: Retrieval-Based Word Learning in Developmental Language Disorder: Verb Learning
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Purdue University (Other)
Collaborators: National Institute on Deafness and Other Communication Disorders (NIDCD) (NIH)
Responsible Party: Principal Investigator, Laurence Leonard, Professor of Speech, Language, & Hearing Sciences, Purdue University
Allocation: Non-Randomized | Model: Factorial | Masking: None | Purpose: Basic Science
Other Study IDs: 1603017480B; R01DC014708 (NIH)
Record Dates: First submitted 2023-08-03; First posted 2023-08-21 (Actual); Results first posted 2025-08-13 (Actual); Last update posted 2025-08-13 (Actual); Status verified 2025-07

CONDITIONS: Developmental Language Disorder; Specific Language Impairment; Language Development
Keywords: word learning; word retrieval; preschool-aged children
MeSH Terms: conditions — Language Development Disorders; Specific Language Disorder

STUDY DESIGN:
Intervention Model Description: Within-participant design in which each child learns words under two conditions.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Children with Developmental Language Disorder (Experimental): These children have a significant delay in language development in the absence of hearing impairment, cognitive delay, autism, or neurological injury/disease.
  Interventions: Behavioral: Retrieval-based verb learning: Repeated Spaced Retrieval condition; Behavioral: Retrieval-based verb learning: Repeated Study condition
- Children with typical language development (Experimental): Children whose language development is as expected for their age.
  Interventions: Behavioral: Retrieval-based verb learning: Repeated Spaced Retrieval condition; Behavioral: Retrieval-based verb learning: Repeated Study condition

INTERVENTIONS:
Behavioral: Retrieval-based verb learning: Repeated Spaced Retrieval condition — A set of novel verbs are practiced on 2 consecutive days (the same verbs are used each day). Half of the novel verbs are learned in the repeated spaced retrieval condition and half are learned in the repeated study condition, with the two conditions interleaved on each day.
  The repeated spaced retrieval condition consists of study and retrieval trials. At the start of the sessions, retrieval trials immediately follow study trials. Thereafter, retrieval trials are spaced for each verb, occurring after 3 other words have intervened between the retrieval trial and the last study trial for that verb.
Behavioral: Retrieval-based verb learning: Repeated Study condition — A set of novel verbs are practiced on 2 consecutive days (the same verbs are used each day). Half of the novel verbs are learned in the repeated spaced retrieval condition and half are learned in the repeated study condition, with the two conditions interleaved on each day.
  The repeated study condition consists of study trials only (with no retrieval practice).

SUMMARY:
Children with developmental language disorder (DLD; also referred to as specific language impairment) experience a significant deficit in language ability that is longstanding and harmful to the children's academic, social, and eventual economic wellbeing. Word learning is one of the principal weaknesses in these children. This project focuses on the word learning abilities of four- and five-year-old children with DLD. The goal of the project is to build on the investigators' previous work to determine whether, as has been found thus far, special benefits accrue when these children must frequently recall newly introduced words during the course of learning. The focus of the current study is verb-learning. The goal of the study is to increase children's absolute levels of verb learning while maintaining the advantage that repeated retrieval holds over comparison methods of learning.

DETAILED DESCRIPTION:
Developmental Language Disorder (DLD) affects language learning in an estimated 7% of children. Although much of the research literature has emphasized difficulties learning grammar, children with DLD also have major deficits in vocabulary. In recent work, the investigators have been examining the benefit of retrieval practice to enhance word learning and retention in preschoolers with DLD. The rationale behind this work is grounded in the growing literature in the field of cognitive psychology which shows that repeated practice in retrieving information results in greater long-term retention than continuous study of that information without opportunities for retrieval. In addition, retrieval practice that occurs after a delay-or "spacing" between study of a word and subsequent recall attempts-can lead to stronger effects.

The investigators have explored the benefits of retrieval practice for preschoolers with DLD and with typical language development (TD), showing that recall and retention for novel words (nouns, adjectives, verbs) were greater when learned using repeated spaced retrieval (RSR) than when learned using repeated study only. Despite benefitting from RSR, children with DLD still showed lower levels of recall than children with TD, in particular in novel verb learning.

In the current study, the investigators seek to improve the absolute levels of word form recall for verbs by modifying the method used previously. Sixteen children with DLD will be recruited for this study along with 16 children with TD matched on chronological age. Using a within-subjects design, children will learn eight novel verbs, four at a time. Each set of four will be learned over two consecutive days, with two words in the RSR condition and two words in a repeated study condition. The referents for these novel words will be video-recorded transitive actions performed by actors on objects and presented on a laptop screen.

In the RSR condition, children will initially hear the word paired with a video of a novel action, immediately be asked to recall the word, and then see/hear it again. After three other words are presented, they will be asked to recall the original word again; this "3" spaced retrieval schedule will continue for the rest of the learning session. In the comparison condition, children will simply hear the words paired with a video of the novel action. In this study, during retrieval practice, children will be prompted to respond with a full sentence containing the verb.

Recall of the verbs will be tested after the learning session on the second day and one week later. At one week, children will also complete a syntactic generalization test in which they are prompted to use the novel verb in a type of sentence that is different from the one used during learning. Finally, children will complete a two-alternative recognition test.

The investigators hypothesize that novel verbs that undergo RSR during the learning period will be learned and recalled better than comparable novel verbs that are assigned to the repeated study condition. This RSR advantage will continue to be observed when the children must use the novel verbs with new actors and objects and will be seen as well in the syntactic generalization test when the children must use the novel verbs in a new sentence frame. Introducing novel verbs representing actions that can be performed on varying objects is expected to improve overall learning. In addition, by having the child produce the verbs in the context of a full sentence, the newly learned verbs should become more integrated with other sentence elements (subjects and direct objects), resulting in a richer representation in memory and consequently, greater recall, recognition, and syntactic flexibility than was observed in the previous novel verb study.

ELIGIBILITY:
Inclusion Criteria:

* a significant deficit in language ability (language test score below cutoff for best sensitivity/specificity) or documented age-appropriate language ability.

normal hearing no evidence of neurological damage or disease scores on tests of nonverbal intelligence above the intellectual disability range not within Autistic range on Autism screening test native English speaker (can be bilingual)

Exclusion Criteria:

* failed hearing screening known neurological damage or disease scores on tests of nonverbal intelligence below the intellectual disability range (standard score less than 75) autism spectrum disorder non-native English speaker

Ages: 48 Months to 71 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 31 (Actual)
Dates: Start 2023-03-01 (Actual); Primary Completion 2024-01-25 (Actual); Study Completion 2024-01-25 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Laurence B. Leonard, PhD, Principal Investigator — Purdue Universtiy
Locations (1):
- Purdue University, West Lafayette, Indiana, United States

IPD SHARING:
Plan to Share IPD: Yes
Data that contribute to our final published results will be made available at www.clinicaltrials.gov.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Data will become available after the results are published or within 12 months from the primary completion date (i.e., the date of final data collection for the primary outcome measure).
Access Criteria: De-identified data will be made publicly available at www.clinicaltrials.gov

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Children with DLD are recruited primarily through speech pathologists and preschool teachers. They are provided with eligibility guidelines and a parent letter. Once the parent is given the letter, they choose to contact us, if interested.
  Children with typical language development are recruited through advertising in preschools.
Pre-assignment Details: Children are initially tested to see if they meet the inclusionary and exclusionary criteria of Developmental Language Disorder. These include falling below age level on a language test, while passing a hearing screening, a non-verbal IQ test, and an autism screener. Many children who are recruited and consented do not meet all these criteria pointing to the fact that DLD is not readily recognizable to non-professionals (parents, preschool teachers).
Period: Overall Study
Arm/Group | Children With Developmental Language Disorder | Children With Typical Language Development
Started | 14 | 17
Completed | 14 | 13
Not Completed | 0 | 4
Not completed — Withdrawal by Subject | 0 | 2
Not completed — Protocol Violation | 0 | 2

BASELINE CHARACTERISTICS:
Population: Baseline population include children who met the inclusionary & exclusionary criteria for Developmental Language Disorder or for Typical Language Development. Those who did not meet the criteria are not included.
Groups:
- Total: Total of all reporting groups
Arm/Group | Children With Developmental Language Disorder | Children With Typical Language Development | Total
Number analyzed (Participants) | 14 | 13 | 27
Age, Continuous [Mean (Standard Deviation); unit: months] | 57.21 (5.19) | 59.00 (5.26) | 58.07 (5.20)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 9 | 7 | 16
  Male | 5 | 6 | 11
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 0 | 1
  Not Hispanic or Latino | 13 | 13 | 26
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 1 | 0 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 2 | 1 | 3
  White | 10 | 11 | 21
  More than one race | 1 | 1 | 2
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 14 | 13 | 27
Maternal Education in Years [Mean (Standard Deviation); unit: years] | 16.71 (3.36) | 17.42 (2.63) | 17.06 (2.89)

OUTCOME MEASURES:

1. Primary Outcome: Verb Recall Accuracy (Number of Verbs Correctly Recalled) in Repeated Spaced Retrieval (RSR) and Repeated Study (RS) Conditions at 5 Mins. for Learned Items
Description: Five minutes after second learning session, child is asked to recall and say the word associated with each novel action learned under each of the two conditions: a condition in which spaced retrieval trials occurred and one in which there were no retrieval trials. For Learned items, each of the four verbs was tested with videos of two of the agent-object pairs the child had seen during the learning period, for a total of 8 recall items. Children were prompted to retrieve/produce the novel verbs in the sentence structure used during learning.
Time Frame: 5 minutes after end of Day 2 (second day) learning period.
Measure: Mean (Standard Error); unit: number of verbs recalled
Arm/Group | Children With Developmental Language Disorder | Children With Typical Language Development
Number analyzed (Participants) | 14 | 13
number of verbs recalled
  Learned 5 min RSR condition | 3.79 (0.60) | 5.31 (0.63)
  Learned 5 min RS condition | 2.86 (0.63) | 3.38 (0.65)
Statistical Analysis 1: Comparison: Children With Developmental Language Disorder; Test type: Superiority; p < 0.0001, LSD test
Statistical Analysis 2: Comparison: Children With Typical Language Development; Test type: Superiority; p < 0.00001, LSD test

2. Primary Outcome: Verb Recall Accuracy (Number of Verbs Correctly Recalled) in Repeated Spaced Retrieval (RSR) and Repeated Study (RS) Conditions at 5 Mins. for Generalized Items
Description: Five minutes after second learning session, child is asked to recall and say the word associated with each novel action learned under one of two conditions: a condition in which spaced retrieval trials occurred and one in which there were no retrieval trials. For Generalized items each of the four verbs was tested with videos of two agent-object pairs that were new (that the child had not seen during the learning period), for a total of 8 recall items. Children were prompted to retrieve/produce the novel verbs in the sentence structure used during learning.
Time Frame: 5 minutes after end of Day 2 (second day) learning period.
Measure: Mean (Standard Error); unit: number of verbs recalled
Arm/Group | Children With Developmental Language Disorder | Children With Typical Language Development
Number analyzed (Participants) | 14 | 13
number of verbs recalled
  Generalized 5 min RSR condition | 3.79 (0.58) | 4.85 (0.60)
  Generalized 5 min RS condition | 2.43 (0.57) | 3.46 (0.59)
Statistical Analysis 1: Comparison: Children With Developmental Language Disorder; Test type: Superiority; p < 0.00001, LSD test
Statistical Analysis 2: Comparison: Children With Typical Language Development; Test type: Superiority; p < 0.00001, LSD test

3. Primary Outcome: Verb Recall Accuracy (Number of Verbs Correctly Recalled) in Repeated Spaced Retrieval (RSR) and Repeated Study (RS) Conditions at 1 Week for Learned Items.
Description: One week after second learning session, child is asked to recall and say the word associated with each novel action learned under one of two conditions: a condition in which spaced retrieval trials occurred and one in which there were no retrieval trials. For Learned items, each of the four verbs was tested with videos of two of the agent-object pairs the child had seen during the learning period, for a total of 8 recall items. Children were prompted to retrieve/produce the novel verbs in the sentence structure used during learning.
Time Frame: 1 week after Day 2 (second day) learning period.
Measure: Mean (Standard Error); unit: number of verbs recalled
Arm/Group | Children With Developmental Language Disorder | Children With Typical Language Development
Number analyzed (Participants) | 14 | 13
number of verbs recalled
  Learned 1 week RSR condition | 3.64 (0.62) | 5.46 (0.64)
  RS condition | 3.50 (0.62) | 3.77 (0.65)
Statistical Analysis 1: Comparison: Children With Developmental Language Disorder; Test type: Superiority; p = 0.78, LSD test
Statistical Analysis 2: Comparison: Children With Typical Language Development; Test type: Superiority; p < .00001, LSD test

4. Primary Outcome: Verb Recall Accuracy (Number of Verbs Correctly Recalled) in Repeated Spaced Retrieval (RSR) and Repeated Study (RS) Conditions at 1 Week for Generalized Items
Description: One week after second learning session, child is asked to recall and say the word associated with each novel action learned under one of two conditions: a condition in which spaced retrieval trials occurred and one in which there were no retrieval trials. For Generalized items, each of the four verbs was tested with videos of two agent-object pairs that were new (that the child had not seen during the learning period), for a total of 8 recall items. Children were prompted to retrieve/produce the novel verbs in the sentence structure used during learning.
Time Frame: 1 week after Day 2 (second day) learning period.
Measure: Mean (Standard Error); unit: number of verbs recalled
Arm/Group | Children With Developmental Language Disorder | Children With Typical Language Development
Number analyzed (Participants) | 14 | 13
number of verbs recalled
  Generalized 1 week RSR condition | 3.57 (0.61) | 5.38 (0.63)
  Generalized 1 week RS condition | 3.57 (0.56) | 3.92 (0.58)
Statistical Analysis 1: Comparison: Children With Developmental Language Disorder; Test type: Superiority; p = 1.00, LSD test
Statistical Analysis 2: Comparison: Children With Typical Language Development; Test type: Superiority; p < 0.00001, LSD test

5. Primary Outcome: Accuracy of Verb Recall (Number of Verbs Correctly Recalled) in a New Structure in Repeated Spaced Retrieval (RSR) and Repeated Study (RS) Conditions
Description: Child is asked to describe the video of a novel action using the novel verb in a frame different from the one learned (i.e.,"X likes to VERB the Y") in repeated spaced retrieval and repeated study conditions. Each verb is tested with four items: three items made use of videos of agent-object pairs the child had seen during the learning period and one item used an agent-object pair that was new. There were eight items total per condition.
Time Frame: 1 week after Day 2 (second day) learning period.
Measure: Mean (Standard Error); unit: number of verbs recalled
Arm/Group | Children With Developmental Language Disorder | Children With Typical Language Development
Number analyzed (Participants) | 14 | 13
number of verbs recalled
  Repeated Spaced Retrieval | 5.29 (1.22) | 10.23 (1.27)
  Repeated Study | 5.57 (1.41) | 7.38 (1.47)
Statistical Analysis 1: Comparison: Children With Developmental Language Disorder; Test type: Superiority; p = 0.75, LSD test
Statistical Analysis 2: Comparison: Children With Typical Language Development; Test type: Superiority; p < 0.01, LSD test

6. Primary Outcome: Verb Recognition (Number of Words Accurately Identified) in Repeated Spaced Retrieval (RSR) and Repeated Study (RS) Conditions for Learned Items.
Description: One week after the learning session, child is asked to indicate (by pointing) which of 2 video options is referred to upon hearing a sentence using a novel word learned in either the repeated spaced retrieval or repeated study condition. Each verb is tested with two items which used videos of agent-object pairs that the child had seen during the learning period, for a total of eight items.
Time Frame: 1 week after Day 2 (second day) learning period.
Measure: Mean (Standard Error); unit: verbs with correct video identified
Groups:
- Children With Developmental Language Disorder: These children have a significant delay in language development in the absence of hearing impairment, cognitive delay, autism, or neurological injury/disease.
  Retrieval-based verb learning: Repeated Spaced Retrieval condition: Novel verbs are practiced on Day 1 using repeated study and retrieval trials. At the start of the session, retrieval trials immediately follow study trials; remaining retrieval trials are spaced for each word (occurring after 3 other words have intervened). This practice schedule is repeated the next day (Day 2).
  Retrieval-based verb learning: Repeated Study condition: Novel verbs are practiced on 2 consecutive days using repeated study trials only, (with no retrieval practice).
- Children With Typical Language Development: Children whose language development is as expected for their age.
  Retrieval-based verb learning: Repeated Spaced Retrieval condition: Novel verbs are practiced on Day 1 using repeated study and retrieval trials. At the start of the session, retrieval trials immediately follow study trials; remaining retrieval trials are spaced for each word (occurring after 3 other words have intervened). This practice schedule is repeated the next day (Day 2).
  Retrieval-based verb learning: Repeated Study condition: Novel verbs are practiced on 2 consecutive days using repeated study trials only, (with no retrieval practice).
Arm/Group | Children With Developmental Language Disorder | Children With Typical Language Development
Number analyzed (Participants) | 14 | 13
verbs with correct video identified
  Learned RSR Condition | 7.00 (0.24) | 7.92 (0.25)
  Learned RS condition | 7.00 (0.24) | 8.00 (0.25)
Statistical Analysis 1: Comparison: Children With Developmental Language Disorder; Test type: Superiority; p < 0.00001, LSD test
Statistical Analysis 2: Comparison: Children With Typical Language Development; Test type: Superiority; p = 0.62, LSD test

7. Primary Outcome: Verb Recognition (Number of Words Accurately Identified) in Repeated Spaced Retrieval (RSR) and Repeated Study (RS) Conditions for Generalized Items.
Description: One week after the learning session, child is asked to indicate (by pointing) which of 2 video options is referred to upon hearing a sentence using a novel word learned in either the repeated spaced retrieval or repeated study condition. Each verb is tested with two items which used videos of agent-object pairs that were new (that the child had not seen during the learning period), for a total of eight items.
Time Frame: 1 week after Day 2 (second day) learning period.
Measure: Mean (Standard Error); unit: verbs wtih correct video identified
Arm/Group | Children With Developmental Language Disorder | Children With Typical Language Development
Number analyzed (Participants) | 14 | 13
verbs wtih correct video identified
  Generalized RSR condition | 7.36 (0.23) | 7.61 (0.24)
  Generalized RS condition | 7.14 (0.23) | 7.77 (0.24)
Statistical Analysis 1: Comparison: Children With Developmental Language Disorder; Test type: Superiority; p = 0.16, LSD test
Statistical Analysis 2: Comparison: Children With Typical Language Development; Test type: Superiority; p = 0.33, LSD test

8. Secondary Outcome: Peabody Picture Vocabulary Test, Fifth Edition
Description: The Peabody Picture Vocabulary is an individually administered, norm-reference test that assesses receptive vocabulary (ability to understand individual words) for children and adults ages 2 years 6 months to 90 years and older. Standard scores are derived from number correct. Standard scores can range from a minimum of 40 and 160. Standard scores between 85 and 115 (1 standard deviation above and below the mean of 100) are interpreted as reflecting receptive vocabulary levels expected for age. Scores below 85 are interpreted as reflecting receptive vocabulary levels below what is expected for age.Scores above 115 are interpreted as reflecting receptive vocabulary levels above what is expected for age.
Time Frame: Test completed at start of study
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Children With Developmental Language Disorder | Children With Typical Language Development
Number analyzed (Participants) | 14 | 13
score on a scale | 98.07 (11.28) | 116.69 (10.98)
Statistical Analysis 1: Comparison: Children With Developmental Language Disorder vs Children With Typical Language Development; Test type: Superiority; p = .54, t-test, 2 sided

9. Secondary Outcome: Maternal Education in Years
Description: Educational attainment of child's mother in terms of years of education
Time Frame: information collected at start of study
Measure: Mean (Standard Deviation); unit: years
Arm/Group | Children With Developmental Language Disorder | Children With Typical Language Development
Number analyzed (Participants) | 14 | 13
years | 16.71 (3.36) | 17.42 (2.36)
Statistical Analysis 1: Comparison: Children With Developmental Language Disorder vs Children With Typical Language Development; Test type: Superiority; p < .001, t-test, 2 sided

ADVERSE EVENTS:
Time Frame: 4 weeks
Arm/Group | Children With Developmental Language Disorder | Children With Typical Language Development
All-Cause Mortality (participants affected / at risk) | 0/14 | 0/13
Serious Adverse Events (participants affected / at risk) | 0/14 | 0/13
Other Adverse Events (participants affected / at risk) | 0/14 | 0/13

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2023-02-24): https://cdn.clinicaltrials.gov/large-docs/66/NCT06001866/Prot_SAP_001.pdf
  • Informed Consent Form (2023-06-07): https://cdn.clinicaltrials.gov/large-docs/66/NCT06001866/ICF_002.pdf